CLINICAL TRIAL: NCT01451658
Title: Endoscopic Treatment Alone Versus Combined Propranolol and Endoscopic Treatment of Acute Variceal Hemorrhage in Patients With Hepatocellular Carcinoma
Brief Title: A Trial of EVL\GVS Alone vs. EVL\GVS Combined Propranolol (S-HCC)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V99C1-026；V100C-024
Record Dates: First submitted 2011-10-10; First posted 2011-10-14 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Gastroesophageal Varices Hemorrhage; Hepatocellular Carcinoma
Keywords: Variceal bleeding; portal hypertension; hepatocellular carcinoma; endoscopic variceal ligation; non-selective beta-blocker; rebleeding
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypertension, Portal | interventions — Propranolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVL or GVS treatment (No Intervention): Endoscopic treatment alone is used for 2nd prevention of gastroesophageal variceal bleeding in patients with HCC.
  endoscopic variceal ligation (EVL) or Gastric Variceal Sclerotherapy (GVS)
- Endoscopic treatment combined propranolol (Experimental): Endoscopic treatment alone versus combined propranolol is used for 2nd prevention of gastroesophageal variceal bleeding in patients with HCC.
  Interventions: Drug: propranolol

INTERVENTIONS:
Drug: propranolol — Starting from 20 mg daily, titrated weekly to decrease heart rate more than 25 % of baseline, administrated during the whole study period
  Other Names: propranolol:Inderal,Cardolol
  Arms: Endoscopic treatment combined propranolol

SUMMARY:
Patients with hepatocellular carcinoma and esophageal varices bleeding were randomized to undergo endoscopic ligation alone (group A) and additive propranolol treatment (group B) after stabilization of their first acute bleeding.

DETAILED DESCRIPTION:
Esophageal variceal bleeding is characteristic of high rebleeding rate and mortality. Thanks to the recent advance of treatment for variceal bleeding such as non-selective beta blocker (NSBB) added to endoscopic ligation further reduce rebleeding in cirrhotic patients, the rebleeding rate and mortality has a marked reduction. However, hepatocellular carcinoma (HCC) is a distinct group characteristic of very poor prognosis in patients with portal hypertension when compared to those of liver cirrhosis only. Therefore, the investigators design a study to randomize patients with HCC and acute variceal bleeding to endoscopic treatment alone and combination with endoscopic treatment and NSBB. This is the two years study.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of HCC
2. endoscopically proven acute variceal bleeding
3. younger than 18 years old or older than 80 years old

Exclusion Criteria:

-Had a terminal illness of any major organ system,such as heart failure, kidney failure,COPD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Rebleeding | 2 year

SECONDARY OUTCOMES:
complication survival | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Veteran General Hospital-Taipei, Taipei, Ming-Chih Hou, MD, Taiwan